CLINICAL TRIAL: NCT01093170
Title: A Phase I Open Label Dose Escalation Trial of RNA-144101 in the Treatment of Geographic Atrophy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was not conducted, no subjects recruited.
Sponsor: Mark Kleinman (Other)
Responsible Party: Sponsor-Investigator, Mark Kleinman, Sponsor/PI, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 144101a
Record Dates: First submitted 2010-03-22; First posted 2010-03-25 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RNA-144101 (Experimental)
  Interventions: Drug: RNA-144101

INTERVENTIONS:
Drug: RNA-144101 — Intravitreous administration of RNA-144101

SUMMARY:
This is a non-randomized, open-label, dose-escalating Phase Ia study performed at a single center designed to evaluate the safety, pharmacokinetics, and preliminary efficacy of intravitreous administration of RNA-144101 in patients with geographic atrophy (GA).

ELIGIBILITY:
Inclusion Criteria:

* Males and females of all races and ethnicities between the ages of 50-99
* Female subjects must be 1-year postmenopausal or surgically sterilized and must have negative serum pregnancy test
* Subjects must have GA from AMD in one or both eyes:
* The study eye will be the eye that meets all inclusion/exclusion criteria
* If both eyes meet criteria, then the eye with the smaller GA lesion will be studied
* If the GA lesions are equal in size, then the eye with the best-corrected visual acuity (BCVA) will chosen as the study eye
* If both eyes have the same lesion size and same BCVA, the right eye will be chosen
* Subjects must have the following GA criteria for inclusion:
* GA lesions with an area > 2.5mm2 and ≤ 20mm2 as determine by fluorescein angiography and fundus autofluorescence
* A clear view to the fundus must be present in order to easily examine the study eye at baseline
* BCVA In the study eye between 20/20 and 20/100 as measured on Snellen chart or 85-50 letters by ETDRS
* Willing and able to provide signed informed consent prior to any study participation

Exclusion Criteria:

* GA due to a disease other than AMD
* Pregnancy or lactation
* Treatment of any systemic infection
* Autofluorescence pattern marked at none, focal or patchy
* Ocular surgery in the study eye in the previous 6 months.
* Presence or history of choroidal neovascularization (wet AMD) in the study eye
* Any inflammatory (autoimmune, uveitis) or neovascular (diabetic retinopathy) disease of the retina
* Any history of glaucoma or disc cupping in the study eye
* Any history of severe dry eye disease
* High myopia > - 8D or high hyperopia > +8D in the study eye
* Presence of life-threatening disease
* Abnormal basal metabolic panel or liver function tests
* Current alcohol or other substance abuse
* Unwilling or unable to provide signed informed consent for any study procedures

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of RNA-144101 as measured by vision testing, ophthalmic and physical exams, vital signs, clinical laboratory testing and AEs. | Through study completion or discontinuation

SECONDARY OUTCOMES:
Pharmacokinetic studies measuring drug concentrations in serum over study period. | Through study completion or discontinuation
Measurement of total aggregate area of GA lesions (as determined by color fundus photography and autofluorescence imaging) | Through duration of study or discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Jayakrishna Ambati, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky / Dept of Ophthalmology, Lexington, Kentucky, United States